CLINICAL TRIAL: NCT06352775
Title: The Effect of Calcium Carbonate on Labor Induction: A Pilot Study
Brief Title: Calcium Carbonate on Labor Induction
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IRB00107112
Record Dates: First submitted 2024-03-07; First posted 2024-04-08 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Pregnancy; Uterine Contraction
Keywords: Pregnancy; Uterine contraction; Calcium carbonate; Labor induction time; Labor dystocia
MeSH Terms: conditions — Dystocia | interventions — Calcium Carbonate

STUDY DESIGN:
Intervention Model Description: The quasi-experimental design will include a prospective treatment group and retrospective historical control group. The prospective treatment group will identify 50 patients who will be voluntarily consented and receive calcium carbonate (500mg every 4 hours, per standardized treatment protocol) plus standard-dose oxytocin. This group will be compared against a retrospective historical control group of 200 randomly selected patients (1:4 ratio) who presented for induction at the same institution within the previous three years and received standard-dose oxytocin alone.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prospective Treatment Group (Experimental): Patients receive calcium carbonate (500mg every 4 hours, per standardized treatment protocol) plus standard-dose oxytocin for labor induction
  Interventions: Dietary Supplement: Calcium Carbonate
- Retrospective Historical Control Group (No Intervention): Patients who presented for induction at the same institution within the previous three years and received standard-dose oxytocin alone for labor induction and were not treated with calcium carbonate

INTERVENTIONS:
Dietary Supplement: Calcium Carbonate — We will be using it in routes and doses consistent with its approved uses. Per the drug label information for Calcium Carbonate USP 500 mg found in the US National Library of Medicine, adults may take 2-4 tablets as symptoms occur and if pregnant to not exceed 10 tablets in 24 hours. Therefore, using a dosing of 500mg every 4 hours will be well below that guidance. When both cervical ripening has been completed and the oxytocin administration begins, the calcium carbonate treatment group will be given calcium carbonate 500mg every 4 hours (not to exceed 10 tablets in 24 hours) until they deliver.
  Arms: Prospective Treatment Group

SUMMARY:
The investigators aim to evaluate the safety and efficacy of administering calcium carbonate to laboring participants undergoing labor inductions. The investigators hypothesize that calcium carbonate is a low-risk preventative measure to decrease oxytocin induction time and dosage, decrease the rate of labor dystocia, decrease the rate of cesarean deliveries, and demonstrate no differences in maternal or neonatal safety outcomes.

DETAILED DESCRIPTION:
The investigators plan to assess (1) duration of induction with oxytocin administration, (2) rate of labor dystocia/failed induction, (3) rate of cesarean section, and (4) maternal/neonatal safety. Currently, calcium carbonate is used by clinicians in patients with varying characteristics, at varying doses, and at various times in their labor process based on their professional preference and experience. The investigators will implement a standardized treatment protocol for calcium carbonate use within a defined patient population who voluntarily agree to prospectively receive the intervention and then analyze predetermined safety and efficacy outcomes in comparison to a historical cohort of patients meeting the criteria for the defined patient population who did not have any documented calcium carbonate use during labor.

ELIGIBILITY:
Inclusion Criteria:

* Adult laboring patients ( ≥ 18 years of age)
* Able to speak and read English or Spanish (for historical cohort, preferred language should be English or Spanish)
* Singleton gestation
* Greater ≥ 37 weeks gestation in vertex presentation
* Present for induction of labor inclusive of medical indication, elective indication at greater than 39 weeks gestation, trial of labor after cesarean
* Receive standard-dose oxytocin during induction

Exclusion Criteria:

* Participants will be excluded from the study if they do not meet the above inclusion criteria or they will be further excluded under the following circumstances:
* Known need for cesarean section prior to induction of labor
* Known allergy to calcium carbonate
* Known contraindication to taking calcium carbonate including renal calculus, high urine calcium levels, elevated serum calcium, low serum phosphate, achlorhydria, or suspected digoxin toxicity.
* Inability to tolerate oral intake (i.e., nausea/vomiting)
* Need to be nothing by mouth (NPO)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Duration of induction time | During the intervention (time from duration of induction with oxytocin start to delivery)
  Participants in the treatment group will have a shorter duration of induction with oxytocin than those in the retrospective historical control group.
Rate of labor dystocia | During the intervention (measured from time of induction to delivery)
  Participants in the treatment group will have a lower rate of labor dystocia than those in the retrospective historical control group.

SECONDARY OUTCOMES:
Rate of cesarean deliveries | During the intervention (measured from time of induction to delivery)
  Participants in the treatment group will have a lower rate of cesarean deliveries than those in the retrospective historical control group.
Total amount of oxytocin after cervical ripening | During the intervention (time on oxytocin after cervical ripening completed to delivery)
  Participants in the treatment group will receive a lower amount of oxytocin than those in the retrospective historical control group.
Gastrointestinal side effects | During the intervention (time on calcium carbonate to delivery)
  Participants in the treatment group will describe gastrointestinal side effects.
Blood loss | Time from delivery to 24 hours of birth
  Participants in the treatment group will experience less blood loss than those in the retrospective historical control group.
Rate of postpartum hemorrhage (>/= 500mL) | Time from delivery to 24 hours of birth
  Participants in the treatment group will experience less postpartum hemorrhage than those in the retrospective historical control group.
Neonatal composite adverse outcomes | Immediately after the birth until the time of discharge, an average of 3 days
  Neonates of participants in the treatment group will have comparable composite adverse outcomes to those born to participants in the retrospective historical control group.

CONTACTS AND LOCATIONS:
Overall Officials: Marie Forgie, DO, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Aurora Sinai Medical Center, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No
Study data will only be shared with those listed on the study team as approved by the internal IRB.